CLINICAL TRIAL: NCT02251314
Title: The Utility and Relevance of Exome Sequence Analysis and Circulating Tumour DNA in Assessing Tumour Heterogeneity in BRAF Mutant Melanoma
Brief Title: Use of Exome Sequence Analysis and Circulating Tumour in Assessing Tumour Heterogeneity in BRAF Mutant Melanoma
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 14-7467
Record Dates: First submitted 2014-09-24; First posted 2014-09-29 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Melanoma
Keywords: BRAF mutant melanoma; circulation tumour DNA; tumour heterogeneity; liquid biopsy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — * Pre-mortem bloods taken to obtain ctDNA
  * Post-mortem bloods and tissue To understand to what extent circulating DNA (found in Blood) represents the genetic content of underlying tumour metastases in BRAF mutant melanoma, and
  * To correlate the appearance of metastasis-specific mutations in the ctDNA with histological features in the tumours such as degree of necrosis, inflammation, microvascular density, and location or size of primary tumour and metastases
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Despite recent advances in cancer treatment, little impact has been made on curing as opposed to controlling cancers over the last several decades. Part of the problem is that investigators have an incomplete understanding of how tumours behave as they evolve and in response to treatment. In this trial, the investigators hope to better understand the evolution of BRAF melanoma in response to drugs a patient may have received such as vemurafenib or dabrafenib. Importantly, the investigators want to understand how the tumours evolve resistance to these drugs and whether this can be predicted through blood tests, in particular of the circulating tumour DNA.

DETAILED DESCRIPTION:
Study population: BRAF mutant melanoma patients

Pre-mortem bloods will be taken from the patient on three occasions at one to thirty days apart from each other, with the first blood draw taking place on the patient's first clinic visit. Six 7 ml EDTA and one 6 ml SST vacutainers of blood (a total of approx. 50 ml of blood) will be taken from the patient.

When death is expected within the next 48-72 hours, the Medical Oncologist/ Radiation Oncologist/ Hematologist OR delegate will revisit the RAP process with the patient and/or family/substitute decision maker to ensure that they are still in agreement. The patient and the families will also be provided with an additional consent form for participation including blood sampling.

ELIGIBILITY:
Inclusion Criteria:

UHN adult patient with BRAF mutant melanoma

Exclusion Criteria:

Non BRAF mutant melanoma patient Pediatric patient Non-UHN patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UHN patients with BRAF mutant melanoma
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2018-04-22 (Actual)

PRIMARY OUTCOMES:
Percentage correlation between circulating tumour DNA and metastatic sites | 3 years

SECONDARY OUTCOMES:
Time to death | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Joshua, Dr., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada